CLINICAL TRIAL: NCT01338818
Title: A 6-month, Open-label Extension to a 40-week, Randomized, Double-blind, Placebo-controlled, Multicenter Efficacy and Safety Study of Methylphenidate Hydrochloride Extended Release in the Treatment of Adult Patients With Childhood-onset ADHD
Brief Title: Open-label Extension Evaluating Methylphenidate Hydrochloride Extended Release in Adults With Attention Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRIT124D2302E1; 2011-000210-19
Record Dates: First submitted 2011-04-15; First posted 2011-04-20 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit /Hyperactivity Disorder,; hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm | interventions — Methylphenidate

ARMS (1):
- Ritalin LA (Experimental): All participants started with Ritalin LA 20 mg/day and increased at weekly intervals in increments of 20 mg/day until reaching the patient's optimal dose 40, 60 or 80 mg/day).
  Interventions: Drug: Ritalin LA (methylphenidate hydrochloride extended release)

INTERVENTIONS:
Drug: Ritalin LA (methylphenidate hydrochloride extended release) — Ritalin LA 20 mg or 30 mg (a racemic mixture of d- and l-thre-Methylphenidate Hydrocloride (MPH), Extended release hard capsules) taken orally once daily in doses of 40, 60, or 80 mg. For 40mg dose patients took (2) Ritalin LA 20mg daily, for 60mg patients took (2) Ritalin LA 30mg daily and for 80mg patients took (2) Ritalin LA 30mg daily + (1) Ritalin LA 20mg daily for their optimal dose.
  Other Names: Ritalin LA, methylphenidate hydrochloride extended release, RIT124D

SUMMARY:
This study will evaluate the long-term safety of methylphenidate hydrochloride extended release in adults with attention deficit/hyperactivity disorder

ELIGIBILITY:
Inclusion Criteria:

1. Completion of the 40-week core study CRIT124D2302 and Week 40 (End of Study) assessments or Patients who meet predefined criteria for treatment failure, were withdrawn from the core study, and have completed core-study week 40 assessments (Premature Discontinuation Visit)

Exclusion Criteria:

1. Patients who, during the core study, developed any psychiatric condition that requires treatment with medication or that may interfere with study participation and /or study assessments.
2. Patients who during the core study developed cardiovascular disorders.
3. Pregnant women.
4. Patients who developed seizures during the core study.
5. Diagnosis of glaucoma, hyperthyroidism, pheochromocytoma.
6. Diagnosis or family history of Tourette's syndrome.
7. Patients who during the core study developed cerebrovascular disorders such as cerebral aneurysm, vascular abnormalities including vasculitis and stroke

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 299 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (15):
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Spring Valley, California
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, West Plam Beach, Florida
  - Novartis Investigative Site, Libertyville, Illinois
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Bellevue, Washington
  - Novartis Investigative Site, Seattle, Washington
- Belgium (5):
  - Novartis Investigative Site, Bruges, Belgium
  - Novartis Investigative Site, Heusden-Zolder, Belgium
  - Novartis Investigative Site, Uccle, Belgium
  - Novartis Investigative Site, Kessel-Lo
  - Novartis Investigative Site, Mechelen
- Colombia (2):
  - Novartis Investigative Site, Santa Fe de Antioquia, Antioquia
  - Novartis Investigative Site, Antioquia
- Novartis Investigative Site, Århus C, Denmark
- Germany (21):
  - Novartis Investigative Site, Bamberg, Germany
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Hamburg, Germany
  - Novartis Investigative Site, Ludwigsburg, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, München, Germany
  - Novartis Investigative Site, Naumburg, Germany
  - Novartis Investigative Site, Nuremberg, Germany
  - Novartis Investigative Site, Wolfsburg, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Landau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Limburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Westerstede/Oldenburg
  - Novartis Investigative Site, Würzburg
- Sweden (2):
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Malmo

REFERENCES:
- [Derived] Boesen K, Paludan-Muller AS, Gotzsche PC, Jorgensen KJ. Extended-release methylphenidate for attention deficit hyperactivity disorder (ADHD) in adults. Cochrane Database Syst Rev. 2022 Feb 24;2(2):CD012857. doi: 10.1002/14651858.CD012857.pub2. PMID 35201607
- [Derived] Ginsberg Y, Arngrim T, Philipsen A, Gandhi P, Chen CW, Kumar V, Huss M. Long-term (1 year) safety and efficacy of methylphenidate modified-release long-acting formulation (MPH-LA) in adults with attention-deficit hyperactivity disorder: a 26-week, flexible-dose, open-label extension to a 40-week, double-blind, randomised, placebo-controlled core study. CNS Drugs. 2014 Oct;28(10):951-62. doi: 10.1007/s40263-014-0180-4. PMID 25183661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Actual enrolment was 299 but one patient entered the extension but did not receive a single dose of the study medication and was subsequently excluded from the All Extension Patients Population
Period: Overall Study
Arm/Group | Ritalin LA
Started | 298
Completed | 262
Not Completed | 36
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 5
Not completed — no longer require study drug | 1
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 4
Not completed — Administrative problems | 3
Not completed — Protocol Deviation | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ritalin LA
Number analyzed (Participants) | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Deaths.
Description: Adverse Events, Serious Adverse Events and Deaths were monitored from week 40 to week 66.
Time Frame: Week 40 - Week 66
Population: All Extension Patients(AEP) analysis set was used for all efficacy and safety analyses of the extension study. AEP was ALL patients who had entered the extension study & received at least 1 dose of Ritalin LA. Enrolment was 299, but 1 pt entered the extension but didn't receive 1 dose of Ritalin LA and was excluded from AEP Population analysis.
Measure: Number; unit: participants
Arm/Group | Ritalin LA
Number analyzed (Participants) | 298
participants
  Adverse Events (Serious and Non Serious) | 208
  Serious Adverse Events | 2
  Deaths | 0

2. Secondary Outcome: Change From Extension Baseline (Week 40) to End of Study (Week 66) in on DSM-IV Attention-Deficit/Hyperactivity Disorder Rating Scale (DSM-IV ADHD RS) Total Score.
Description: Attention-Deficit/Hyperactivity Disorder Rating Scale (DSM-IV ADHD RS) total score consists of 18 items directly adapted from the ADHD symptom list according to the DSM-IV. The DSM-IV ADHD RS total score was calculated as the sum of the Inattentive and the Hyperactive-Impulsive subscores. The 18 items are rated from 0 ("rarely or never") to 3 ("Very often"). The total score ranges from 0 to 54. Decrease in the DSM-IV ADHD RS total score indicates improvement, therefore a greater decrease (change at Final Visit compared to baseline) indicates a greater improvement in ADHD symptoms. Last Observation Carried Forward (LOCF) applied for each patient with data in extension period. If no post-baseline is available, it is considered as missing.
Time Frame: week 40 - week 66
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ritalin LA
Number analyzed (Participants) | 298
scores on a scale | -7.2 (11.00)

3. Secondary Outcome: Change From Extension Baseline (Week 40) to End of Study (Week 66) on Sheehan Disability Scale (SDS) Total Score
Description: SDS,5-self-rated questionnaire to measure the extent a pt's disability due to an illness/health problem interferes with work/school,social life/leisure,family life/home. First 3 items, pts are asked how their symptoms disrupted their regular activities over the past 7d in each using a scale from 0(not at all)-10(extremely) Each subscale(work disability, social life disability, family life disability)can be scored independently or combined into a total score(sum of the non-missing responses for items 1-3)from 0-30,higher scores indicate significant functional impairment. Subscale scores>5 suggest impairment in that subscale area. Final 2 items ask pts about the # of days their symptoms caused them to miss school/work and # of days their symptoms caused them to be underproductive at school/work.(These items were not included in the total score.) Before responding to SDS items 1-3, pts were verbally instructed to recall the past 7d, items 4-5 refer to the last week w/in the item wording.
Time Frame: week 40 - week 66
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ritalin LA
Number analyzed (Participants) | 298
Scores on a scale | -4.8 (6.88)

ADVERSE EVENTS:
Arm/Group | Ritalin LA
Serious Adverse Events (participants affected / at risk) | 2/298
Other Adverse Events (participants affected / at risk) | 163/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ritalin LA (N=298)
Pancreatitis (Gastrointestinal disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ritalin LA (N=298)
Palpitations (Cardiac disorders) | 6
Tachycardia (Cardiac disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 9
Gastroenteritis (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 57
Sinusitis (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 14
Weight decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 23
Headache (Nervous system disorders) | 42
Agitation (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 11
Depressed mood (Psychiatric disorders) | 6
Initial insomnia (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 11
Sleep disorder (Psychiatric disorders) | 7
Dysmenorrhoea (Reproductive system and breast disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.